CLINICAL TRIAL: NCT07220369
Title: Evaluation of Ingestible Mini-pill for Gastrointestinal Regional Luminal Content Sampling
Brief Title: Gut Mini-Pill Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Principal Investigator, Alice Lichtenstein, Director of Cardiovascular Research Team, Tufts University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Device Feasibility
Other Study IDs: 5011
Record Dates: First submitted 2025-10-01; First posted 2025-10-23 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Gut Microbiota
Keywords: gut; mini-pill; gut sampling; gut microbiota

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plant-based meat alternative entree (Experimental): Entree that is composed of a plant-based meat alternative
  Interventions: Other: plant-based meat alternative entrees; Device: mini-pill
- meat entree (Experimental): entree that is composed of meat
  Interventions: Device: mini-pill; Other: meat based entree

INTERVENTIONS:
Other: plant-based meat alternative entrees — 2 plant-based meat alternatives per day
  Arms: Plant-based meat alternative entree
Device: mini-pill — mini-pills which sample at different locations in the gut
Other: meat based entree — 2 meat based entrees per day
  Arms: meat entree

SUMMARY:
The purpose of this proof-of-concept study in humans is to determine if a noninvasive, ingestible device, called a "mini-pill", can collect gastrointestinal (GI) luminal content samples from 2 different locations along the GI tract after consumption of diets differing in protein source (meat and plant-based meat alternatives). The mini-pills will be recovered in the stool. We will analyze the microbial profile of the mini-pill contents and in stool, and also measure blood biomarkers related to cardiometabolic risk, to better understand the relationship between diet, microbiota and health.

DETAILED DESCRIPTION:
The ingestible mini-pill is a non-invasive, single-use, passive collection device that is not intended for diagnosis or treatment. The mini-pills have already been developed, tested and validated by two Tufts researchers, Drs. Sameer Sonkusale (School of Engineering) and Giovanni Widmer (School of Veterinary Medicine), in vitro, ex vitro, and in vivo in animal models (Supplement 1: Research Strategy and Supplement 2: Soft Autonomous Ingestible Device for Sampling the Small Intestinal Microbiome, Del-Rio-Ruiz R et al., manuscript in review). A NSR device designation is being sought from the IRB to conduct a 2-phase randomized-controlled double blind crossover trial in humans by providing two entrées per day containing either meat or plant-based meat alternatives for up to 3 weeks each. After 2 weeks on each diet, participants will consume a provided breakfast meal and then be asked to swallow 6 mini-pills along with a blue food coloring dissolved in 50 mL of water, return home and collect stool samples until all the mini-pills are recovered (varies between 2 and 4 days, but can be up to 6 days). This protocol will allow us to describe the diet-induced progressive change in the GI tract microbiota prior to and including that in the stool.

ELIGIBILITY:
Inclusion Criteria:

* Men and postmenopausal women
* Age >50 to <75 years
* BMI >20 to <35 kg/m2
* Normotensive with or without medication
* Normal gastrointestinal function with regular bowel movements at least once every other day
* Normal kidney and liver function
* Willingness to swallow the mini-pills
* Willingness to collect and return multiple stool samples
* Adequate refrigerator and freezer space to store study entrées
* Intent to remain in the greater Boston area during the intervention periods

Exclusion Criteria:

* Individuals self-reporting adhering to any type of vegetarian diet
* Lack of willingness to restrict fish intake to less than once per week during the dietary intervention phases
* Allergy/intolerance/religious reasons to avoid study foods or food ingredients, including known hypersensitivity to Blue 1 food coloring and wheat gluten.
* Regular use of prebiotics or probiotics within the past 3 months
* Regular use of laxatives or fiber supplements
* Chronic constipation
* Chronic use of antibiotics (except topical)
* Regular use of stomach acid lowering and weight loss medications such as GLP-1 agonists
* Use of dental prophylaxis
* Planned colonoscopy 2 months prior to or during the study period
* Gastroparesis
* Swallowing disorder, or inability or difficulty taking pills
* Malabsorptive and inflammatory bowel disease, diverticulosis, and history of diverticulitis, gastric/ esophageal/intestinal surgery, including lap banding or bariatric surgery.
* History of bowel obstruction, pancreas and liver disorders.
* Any form of active substance abuse or dependence (including drug or alcohol abuse). This information will be stored in REDCAP in a subsection that has no identifiers.
* Established major chronic diseases such as cardiovascular disease, diabetes, active cancer within the last 5 years, or any significant medical condition at the study MD's discretion
* A clinical condition that, in the judgment of the study MD or principal investigator, could potentially pose a health risk to the subject while involved in the study.
* Unwillingness to adhere to study protocol
* Intent to increase or decrease body weight during the study period
* No Social Security number (for payment and IRS forms).
* Individuals who directly report to any member of the research team.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Test feasibility of the mini-pill to characterize differential changes inducted by a meat-rich and plant-based meat alternative-rich diet on the gut microbial profile | 8 weeks
  Using luminal content collected by the gut mini-pill to compare the microbiome and metabolome after subjects consumed a meat-rich and plant-based meat alternative-rich diet

SECONDARY OUTCOMES:
Test feasibility of the mini-pill to characterize differential changes inducted by a meat-rich and plant-based meat alternative-rich diet on cardiometabolic risk factors | 8 weeks
  Using luminal content collected by the gut mini-pill to compare the cardiometabolic after subjects consumed a meat-rich and plant-based meat alternative-rich diet

CONTACTS AND LOCATIONS:
Overall Officials: Alice H Lichtenstein, D.Sc., Principal Investigator — Tufts University
Locations (1):
- Jean Mayer Human Nutrition Research Center on Aging, Boston, Massachusetts, United States

DOCUMENTS (1):
  • Study Protocol (2024-05-28): https://cdn.clinicaltrials.gov/large-docs/69/NCT07220369/Prot_000.pdf